CLINICAL TRIAL: NCT05945771
Title: Effects of Acute Grape Seed Extract Supplementation on Muscle Metaboreflex in Healthy
Brief Title: Effects of Acute Grape Seed Extract Supplementation on Muscle Metaboreflex in Healthy Young Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 107-2122-EXP
Record Dates: First submitted 2023-07-03; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Dietary Supplementation
MeSH Terms: interventions — Grape Seed Extract

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized double blind grape seed extract design (Active Comparator): Grape seed extract
  Interventions: Dietary Supplement: Grape seed extract
- Control (Placebo Comparator): Placebo (starch)
  Interventions: Dietary Supplement: Grape seed extract

INTERVENTIONS:
Dietary Supplement: Grape seed extract — Acute effect of dietary supplementation with GSE on hemodynamic responses during static exercise and muscle metaboreflex and during cycling exercise.

SUMMARY:
The aim of this study was to determine whether grape seed extract (GSE) supplementation could reduce the blood pressure (BP) in response to static exercise and post exercise muscular ischemia (PEMI) in normotensive young adults. In 12 healthy subjects (7 male and 5 female, 24.6±3.4 yr), we compared acute effect of both GSE (600 mg) and placebo (PL: 600 mg) on changes from rest in systolic BP (SBP), diastolic BP (DBP), mean arterial pressure (MAP), heart rate (HR), stroke volume (SV), cardiac output (CO), and total peripheral resistance (TPR) during static exercise (SE) and PEMI. Subjects completed 2 min of SE at 30% of maximal voluntary contraction (MVC) followed by 2 min of PEMI.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers (SBP < 120 mmHg, DBP < 80 mmHg)

Exclusion Criteria:

* cardiovascular and/or pulmonary disease,
* musculoskeletal disorders
* medications that prevent the safe completion of the exercise protocol

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2022-05-01 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Systolic blood pressure (mmHg) by sphygmomanometer | 24 hours
  Measured from the brachial artery
Diastolic blood pressure (mmHg) by sphygmomanometer | 24 hours
  Measured from the brachial artery
Mean arterial pressure (mmHg) | 24 hours
  calculated (MAP = (SBP-DBP)/3 + DBP
Heart rate (bpm) | 24 hours
  measured using Physio Flow (non-invasive device)
Stroke volume (ml) | 24 hours
  measured using Physio Flow (non-invasive device)
Cardiac output (l/min) | 24 hours
  calculated: HR (bpm) x SV (ml)
Total peripheral resistance (mmHg/l/min) | 24 hours
  calculated: MAP (mmHg) / CO (l/min)

CONTACTS AND LOCATIONS:
Overall Officials: Jong-Kyung Kim, Principal Investigator — California Baptist University
Locations (1):
- California Baptist University, Riverside, California, United States

IPD SHARING:
Plan to Share IPD: Undecided